CLINICAL TRIAL: NCT06531044
Title: Relationship Between Gross Motor Coordination and Balance in Children With Spastic Cerebral Palsy
Acronym: CP
Status: Recruiting | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Alaa Noureldeen Kora, Lecturer, Sinai University
Other Study IDs: P.T.REC/012/005131
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Balance; Gross Motor Coordination
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 of children with cerebral palsy: Children with spastic cerebral palsy will be enrolled in this study upon fulfilling the following inclusion criteria: They were scored Level I on the Gross Motor Function Classification System (GMFCS).

SUMMARY:
This study aims to determine if there is a connection between gross motor coordination and balance in children with spastic cerebral palsy. Since these children often struggle with balance and other motor skills, researchers hypothesize that there is no link between the two abilities.

DETAILED DESCRIPTION:
PURPOSE:

To examine the relationship between the gross motor coordination and balance in children with spastic cerebral palsy.

BACKGROUND:

Motor coordination is required for the effective acquisition of movements and effortless performance. Gross motor coordination involves numerous skills, including balance, bilateral movement, agility, and speed. Children with cerebral palsy exhibit a deterioration in gross motor coordination ability.

The lack of postural control in children with cerebral palsy impairs functional balance. According to studies, children with cerebral palsy have poorer static and dynamic balance responses than typically developing children.

HYPOTHESES:

- There is no relationship between gross motor coordination and balance in children with spastic cerebral palsy.

RESEARCH QUESTION:

- Is there a relationship between gross motor coordination and balance in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. They were scored Level I on the Gross Motor Function Classification System (GMFCS).
2. The subjects' age was from five to eleven years.
3. They were at least 1-meter-tall and not less 20 Kg.
4. They had to comprehend verbal commands.
5. They were score 1 to 1+ based on Modified Ashworth' Scale.

Exclusion Criteria:

1. Contracture, deformity and/or tightness in upper or lower limbs.
2. Botulinum toxin in the last year.
3. Recent fracture.
4. Vertigo or dizziness.
5. Epilepsy.
6. Osteoporosis.
7. Recent operation in the six months at least (according to the type of operation).

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with spastic cerebral palsy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
balance. | 1 day - one session
  Biodex Balance System will be used to assess balance.
gross motor coordination. | 1 day - one session
  - Gross Motor - BOT -2 will be used to assess gross motor coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Sharing Individual Patient Data (IPD) is often hindered by privacy concerns, data security risks, legal and ethical obligations, resource limitations, and data quality issues.